CLINICAL TRIAL: NCT05791162
Title: Interest of Follicular Helper Lymphocytes / Regulatory Follicular Helper Lymphocytes Ratio to Characterize and Predict Poor Prognosis Forms in IgA Nephropathy: an Exploratory Proof-of-concept Study
Brief Title: Interest of Follicular Helper Lymphocytes / Regulatory Follicular Helper Lymphocytes Ratio in IgA Nephropathy
Acronym: LYMFONI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/748
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Glomerulonephritis, IGA
Keywords: Follicular helper T cells; Follicular regulatory T cells
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IgA nephropathy in follow-up (arm 1) (Other): Diagnosis of IgA nephropathy from 2009, with a minimum follow-up for nephropathy of 5 years
  Interventions: Other: Blood collection; Other: Urine sample
- Newly diagnosed IgA nephropathy (arm 2) (Other): Diagnosis of IgA nephropathy during the study period
  Interventions: Other: Blood collection; Other: Urine sample
- CD163s control (arm 3) (Other): Diagnosis of Lupus or ANCA-associated vasculitis or polycystic kidney disease
  Interventions: Other: Urine sample

INTERVENTIONS:
Other: Blood collection — Collection of 3 blood tubes at inclusion and relapse (arm 1) or at inclusion, initiation of treatment and at 3 and 6 months post-diagnosis (arm 2)
  Arms: IgA nephropathy in follow-up (arm 1); Newly diagnosed IgA nephropathy (arm 2)
Other: Urine sample — Collection of 20 cc of urine at inclusion and relapse (arm 1) or at inclusion, initiation of treatment and at 3 and 6 months post-diagnosis (arm 2) or at inclusion only (arm 3)

SUMMARY:
This study aims to investigate the relevance of the Tfh/Tfr (Follicular helper T cells/ Follicular regulatory T cells) ratio in patients with IgA nephropathy:

* To identify a differential expression of the Tfh/Tfr ratio in patients considered stable or progressive
* To predict, at diagnosis, the clinical evolution of the disease (progressive or stable form) in the first year.

ELIGIBILITY:
Inclusion Criteria:

* IgA nephropathy histologically proven on renal biopsy according to KDIGO criteria, with 8 permeable glomeruli (patients diagnosed from 2009 with a minimum follow-up for their nephropathy of 5 years (arm 1) or patients diagnosed during the study (arm 2))

Control patients: Lupus or ANCA-associated vasculitis or polycystic kidney disease (arm 3)

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subjects with no social security coverage.
* Pregnancy / No effective contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Form of IgA nephropathy exhibited by the patient (progressive or stable) | 12 months
  Patient with a diagnosis before the start of the study: IgA nephropathy with a GFR of less than 45 ml/min/1.73 m2 and/or proteinuria >0.5 g/day and/or hematuria (microscopic or macroscopic) will be considered progressive.
  Patient with diagnosis during the study: will be considered as progressive an IgA nephropathy for which the GFR will decrease compared to the inclusion (diagnosis) of more than 5 ml/min/1.73 m2 and/or with a proteinuria >0.5 g/day and/or with a microscopic hematuria on at least one of the samples carried out in a period of one year after the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Melchior Chabannes, MD, Principal Investigator — Nephrology, CHU Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France